CLINICAL TRIAL: NCT00440076
Title: Phase II Study of PS341 (VELCADE) in Myelodysplastic Syndromes (MDS). EudraCT Number 2004-002935-23
Brief Title: Velcade in Myelodysplastic Syndrome - Pilot Study
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDS0104
Record Dates: First submitted 2007-02-23; First posted 2007-02-26 (Estimated); Last update posted 2015-04-23 (Estimated); Status verified 2015-04

CONDITIONS: MDS
Keywords: MDS; Velcade
MeSH Terms: interventions — Bortezomib

INTERVENTIONS:
Drug: Velcade

SUMMARY:
This is a four-center open-label study designed to determine activity of Velcade in Myelodysplastic Syndrome (MDS) patients. A total of 28 subjects will be enrolled. The patients will be registered to GIMEMA Data Center before therapy starts and after inclusion criteria verification.

DETAILED DESCRIPTION:
The Myelodysplastic Syndromes (MDS) are an heterogeneous group of clonal disorders of the hematopoietic stem cell characterized by ineffective hematopoiesis leading to peripheral cytopenias, and variable risk of progression to more advanced disease and/or transformation to acute myeloid leukemia (AML). The disease affects predominantly elderly individuals (median age 69 years); the overall incidence is about 4 per 100,000 individuals but this rises to > 30 per 100,000 in the over 70 year age population.

Therapy for MDS has included hematopoietic growth factors (in primis EPO, in combination or not with granulocyte-colony stimulating factor- G-CSF or granulocyte-colony stimulating factor-GM-CSF), differentiating agents, immunotherapy, low dose chemotherapy strategies, AML-like induction regimens, traditional cytotoxic agents, and hematopoietic stem cell transplantation (HSCT) strategies. With the exception of HSCT, which can result in long-term survival in 23% to 50% of patients (Ref. 10) therapy for MDS has not consistently shown a survival advantage, and also modest results have been obtained in an attempt to improve anemia and/or the other cytopenias, and to decrease the number of red blood cell (RBC) transfusions. Furthermore, MDS is primarily a disease of older patients who cannot tolerate aggressive therapy and therefore cannot receive HSCT.

No therapy has thus been considered standard for MDS, and supportive therapy, including RBC transfusions, platelet transfusions and antibiotic therapy has often been focus of care, especially in the older patient population.

VELCADE™ (bortezomib) for injection is a small molecule proteasome inhibitor developed by Millennium Pharmaceuticals, Inc., (MPI) as a novel agent to treat human malignancies. VELCADE is currently approved by the US FDA for the treatment of multiple myeloma patients who have received at least 2 prior therapies and have demonstrated disease progression on the last therapy. VELCADE is a modified dipeptidyl boronic acid derived from leucine and phenylalanine; its chemical name is N pyrazinecarbonyl L phenylalanine L leucine boronic acid and has a molecular weight of 384.25 daltons.

Data from non clinical and clinical studies conducted to date support the development of Velcade for the treatment of human malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 -75 years.
* Patients with the following clinical diagnosis: RA(FAB) or RCMD (WHO), RARS (FAB) or RCDM-RS(WHO), RAEB (FAB) or RAEB I (WHO), RAEB II (WHO), and:

  * IPSS intermediate-2 (score 1.5-2) or high (score 2.5-3) not previously treated with chemotherapy (CT) and not eligible for intensive chemotherapy or allogeneic stem cell transplantation (SCT), or
  * IPSS intermediate-1(score 0.5-1) or low (score 0), EPO or immunosuppressive (Cyclosporine, CSA; anti-tymocyte globulin, ATG) therapies resistant or not eligible for these therapies, and transfusion dependent.
* Patients willing and able to comply with the protocol requirements.
* Patients given voluntary written informed consent to participate in the study, with the understanding that consent may be withdrawn at any time without prejudice to future medical care.
* Male and female patients willing to use acceptable methods for contraception, for the duration of the study.
* Patients with WHO performance Status (PS) 0-2, and life expectancy > 3 months.
* Renal function tests ≤ 2 x upper limit of normal values.
* AST/GOT, ALT/GPT ≤ 2.5 x upper limit of normal values.
* Total bilirubine ≤ 1.5 x upper limit of normal value.

Exclusion Criteria:

* Patient has Grade 2 (as defined by the NCI Common Toxicity Criteria-CTC) peripheral neuropathy within 14 days before enrollment.
* Patient has hypersensitivity to bortezomib, boron or mannitol.
* Patient has received prior treatment with bortezomib
* Patient is pregnant or nursing
* Patient has received other investigational drugs within 14 days before enrollment
* Patient has received prior chemotherapy
* Patient had a major surgery within 4 weeks before enrollment
* Patient had myocardial infarction within 6 months of enrollment or has class III-IV heart failure, uncontrolled angina or arrhythmias
* Patient has been treated for previous malignancy within 5 years before enrollment
* Patient has uncontrolled hypertension or diabetes mellitus
* Patient is known to have HBV or HCV active hepatitis or is human immunodeficiency virus (HIV)-positive
* Patient has systemic infections requiring treatment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2006-08; Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
to determine activity of Velcade in patients with MDS, intermediate-2 or high risk, and intermediate-1 or low risk unresponsive or not eligible for treatment with erythropoietin or immunosuppressive agents as assessed according to response criteria.

SECONDARY OUTCOMES:
to determine whether Velcade prolongs time to progression and/or survival; safety and tolerability as assessed by incidence of clinical and laboratory toxicities; quality of life in relation to neurotoxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Giuliana ALIMENA, MD, PHD, Principal Investigator — Università degli Studi di Roma "La Sapienza", Dipartimento di Biotecnologie Cellulari ed Ematolgia
Locations (4):
- Italy (4):
  - Istituto di Ematologia e Oncologia Medica L. e A. Seragnoli, Bologna, Bologna
  - Ospedale Niguarda "Ca Grande", Milan, Milano
  - Centro Oncologico Basilicata, Rionero in Vulture, Potenza
  - A.O Umberto I, Roma, Roma